CLINICAL TRIAL: NCT03882359
Title: MVT-100: Advancing the Clinical Use of Perflutren Ultrasound Contrast Agents for Suboptimal Echocardiograms
Brief Title: An Ascending Dose Comparison of MVT-100 to Definity in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Microvascular Therapeutics, LLC (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 00029941; 1R44HL137447-01A1 (NIH)
Record Dates: First submitted 2019-02-15; First posted 2019-03-20 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Heart Diseases
Keywords: echo; echocardiogram; Healthy Volunteers; Definity
MeSH Terms: conditions — Heart Diseases | interventions — Echocardiography; perflutren

STUDY DESIGN:
Intervention Model Description: Ascending dose comparison in healthy volunteers
Who Masked: Outcomes Assessor
Masking Description: The interpreter of echocardiograms in the trial is blinded to the drug which was administered, MVT-100 or Definity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Definity (Active Comparator): Each subject receives 100 uL x 2, 200 uL x 3, 300 uL x 2 or 1 vial of DEFINITY® 100 diluted in 50 mL of NS as follows: Two milliliter bolus over 10 seconds prior to each infusion rate;, then infusions will run for 5 minutes at 60 mL per hour, 5 minutes at 90 mL per hour, 5 minutes at 100 mL per hour and 5 minutes at 120 mL per hour.
  Interventions: Diagnostic Test: Echocardiogram; Drug: Definity
- MVT-100 (Experimental): Each subject receives 100 uL x 2, 200 uL x 3, 300 uL x 2 or 1 vial of MVT-100 diluted in 50 mL of NS as follows: Two milliliter bolus over 10 seconds prior to each infusion rate;, then infusions will run for 5 minutes at 60 mL per hour, 5 minutes at 90 mL per hour, 5 minutes at 100 mL per hour and 5 minutes at 120 mL per hour.
  Interventions: Diagnostic Test: Echocardiogram; Drug: MVT-100

INTERVENTIONS:
Diagnostic Test: Echocardiogram — Images will be recorded in parasternal long, short axis, apical four, two, and three chamber views according to the American Society of Echocardiography (ASE) 17 segment model. Each assessment will include one round of low MI imaging (<0.3) and one round of very low MI imaging (<0.2) in each of the pre-specified windows according to the 2014 ASE Sonographer Guidelines.
  A baseline echocardiogram will be performed prior to the administration of DEFINITY® or MVT-100. Assessments will be made three times, once from 0 - 1 ½ minutes following injection, once between 1 ½ minutes to 3 minutes following IV injection and once from 3 - 4 ½ minutes following IV injection. Assessments at each time point will include one round of low MI imaging (<0.3) and one round of very low MI imaging (<0.2). Each round will include the views in the following order: parasternal long, parasternal short, apical 4, apical 2 and apical 3.
Drug: MVT-100 — After randomization, MVT-100, the experimental drug, is administered via IV infusion or bolus administration and echocardiograms are subsequently obtained.
  Arms: MVT-100
Drug: Definity — After randomization, Definity, the active comparator, is administered via IV infusion or bolus administration and echocardiograms are subsequently obtained.
  Arms: Definity

SUMMARY:
Definity (perflutren lipid microspheres, Lantheus Medical Imaging) is an ultrasound contrast indicated for use in patients with suboptimal echocardiograms to opacify the left ventricular chamber and to improve the delineation of the left ventricular endocardial border. MVT-100 (the investigational pharmaceutical) is similar to Definity, with the exception of the removal of one lipid in the lipid blend and substitution of another lipid. This study is intended to evaluate the safety and efficacy of MVT-100 using a single ascending dose design in healthy volunteers. Patients are randomized to receive either MVT-100 or Definity and undergo echocardiograms after receiving either MVT-100 or Definity via bolus or IV infusion administration. The primary endpoints evaluated are safety and endocardial border delineation.

DETAILED DESCRIPTION:
Ultrasound is one of the most common imaging examinations and has advantages of absence of ionizing radiation, portability and relatively low cost. Ultrasound contrast agents are used to improve the accuracy of ultrasound and Definity (perflutren) is the world's leading ultrasound contrast agent but perflutren has to be refrigerated and has a side effect of back pain. The investigators have developed a new, improved perflutren, MVT-100, with potential for room temperature storage.

Ultrasound contrast agents are used to increase the backscatter (signal intensity of blood vessels and tissues to improve diagnostic accuracy) of ultrasound imaging. In the US ultrasound contrast agents are FDA approved for echocardiography to improve endomyocardial border definition.

MVT-100 reflects the ultrasound to provide strong back-scattering. MVT-100 microbubbles resonate with ultrasound to provide strong harmonic signals. MVT-100 microbubbles will cavitate with higher levels of ultrasound and cavitation may be stable or inertial depending upon acoustic parameters and other factors.

The study is a multi centre ascending dose comparison of Definity and MVT-100 for use in echocardiography and will be performed in a sample of healthy volunteers who are randomized to receive either Definity or MVT-100.

This trial will assess safety and evaluate the following imaging metrics:

* Determine the optimal dose of MVT-100 by comparing MVT-100 vs Definity in the change from baseline of quantitative left ventricular opacification
* Evaluation of qualitative left ventricular opacification (LVO)
* Evaluation of endocardial border delineation
* Evaluation of endocardial border length
* Evaluation of duration of useful contrast

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 19 years of age or older, male or female
* Female subjects must no longer have child-bearing potential (>1-year post menopause or surgically sterilized), or must

  * have a negative urine pregnancy test, and
  * be using and continue to use for 30 days after the study a medically effective method of contraception
* Adequate hematologic, renal and hepatic function, as defined by:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Hemoglobin ≥ 90 g/L
* Plasma creatinine< 1.5 x ULN
* Total bilirubin within normal limits (< 2.5 x ULN if Gilbert's syndrome)
* Aspartate transaminase (AST) and Alanine transaminase (ALT) < 2.5 x ULN
* Subject must be willing and able to understand the study and provide written Informed Consent to participate in the study

Exclusion Criteria:

* Myocardial infarction within six months prior to enrollment
* Unstable angina, NYHA Class II or greater congestive heart failure
* EKG evidence of uncontrolled arrhythmia or history of clinically significant arrhythmia within the past six months
* Clinically significant Chronic Obstructive Pulmonary Disease (COPD) or other pulmonary condition that is not controlled by medication or requires oxygen frequently or continuously
* A history of pulmonary emboli
* Known hypersensitivity to perflutren, DEFINITY® or other echo contrast agent
* Inability to remain supine for 60 minutes
* Oxygen saturation < 95% on room air
* History of allergic reaction attributed to compounds of similar chemical composition to MVT-100 or DEFINITY® or soy or egg allergies (see Investigator's Brochure)
* Subject has received any investigational drug within thirty (30) days prior to enrollment into the study
* Inability to comply with study procedures
* Subjects with any medical condition deemed by the investigator to make the subject inappropriate for participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
QT Interval | Day of study
  The null hypothesis for safety (H0) will be: MVT-100 is not as safe as DEFINITY®. The alternative hypothesis (HA) for safety will be: MVT-100 is equivalent to, or safer than, DEFINITY®. Specifically, the following hypotheses will be tested:
  HA: Δ2min QT interval EKG(MVT-100) ≤ Δ2min QT interval EKG(Definity®) HA: Δ2min Blood Pressure(MVT-100) ≤ Δ2min Blood Pressure(Definity®) HA: Δ2min Heart Rate(MVT-100) ≤ Δ2min Heart Rate(Definity®) HA: Δ2min O2(MVT-100) ≤ Δ2min O2(Definity®) HA: Other Symptom(2min post MVT-100) ≤ Other Symptom(2min post Definity®)
Blood Pressure | Day of study
  The null hypothesis for safety (H0) will be: MVT-100 is not as safe as DEFINITY®. The alternative hypothesis (HA) for safety will be: MVT-100 is equivalent to, or safer than, DEFINITY®. Specifically, the following hypotheses will be tested:
  HA: Δ2min QT interval EKG(MVT-100) ≤ Δ2min QT interval EKG(Definity®) HA: Δ2min Blood Pressure(MVT-100) ≤ Δ2min Blood Pressure(Definity®) HA: Δ2min Heart Rate(MVT-100) ≤ Δ2min Heart Rate(Definity®) HA: Δ2min O2(MVT-100) ≤ Δ2min O2(Definity®) HA: Other Symptom(2min post MVT-100) ≤ Other Symptom(2min post Definity®)
Heart Rate | Day of study
  The null hypothesis for safety (H0) will be: MVT-100 is not as safe as DEFINITY®. The alternative hypothesis (HA) for safety will be: MVT-100 is equivalent to, or safer than, DEFINITY®. Specifically, the following hypotheses will be tested:
  HA: Δ2min QT interval EKG(MVT-100) ≤ Δ2min QT interval EKG(Definity®) HA: Δ2min Blood Pressure(MVT-100) ≤ Δ2min Blood Pressure(Definity®) HA: Δ2min Heart Rate(MVT-100) ≤ Δ2min Heart Rate(Definity®) HA: Δ2min O2(MVT-100) ≤ Δ2min O2(Definity®) HA: Other Symptom(2min post MVT-100) ≤ Other Symptom(2min post Definity®)
Oxygen Saturation | Day of study
  The null hypothesis for safety (H0) will be: MVT-100 is not as safe as DEFINITY®. The alternative hypothesis (HA) for safety will be: MVT-100 is equivalent to, or safer than, DEFINITY®. Specifically, the following hypotheses will be tested:
  HA: Δ2min QT interval EKG(MVT-100) ≤ Δ2min QT interval EKG(Definity®) HA: Δ2min Blood Pressure(MVT-100) ≤ Δ2min Blood Pressure(Definity®) HA: Δ2min Heart Rate(MVT-100) ≤ Δ2min Heart Rate(Definity®) HA: Δ2min O2(MVT-100) ≤ Δ2min O2(Definity®) HA: Other Symptom(2min post MVT-100) ≤ Other Symptom(2min post Definity®)
Other Symptoms | Day of study
  The null hypothesis for safety (H0) will be: MVT-100 is not as safe as DEFINITY®. The alternative hypothesis (HA) for safety will be: MVT-100 is equivalent to, or safer than, DEFINITY®. Specifically, the following hypotheses will be tested:
  HA: Δ2min QT interval EKG(MVT-100) ≤ Δ2min QT interval EKG(Definity®) HA: Δ2min Blood Pressure(MVT-100) ≤ Δ2min Blood Pressure(Definity®) HA: Δ2min Heart Rate(MVT-100) ≤ Δ2min Heart Rate(Definity®) HA: Δ2min O2(MVT-100) ≤ Δ2min O2(Definity®) HA: Other Symptom(2min post MVT-100) ≤ Other Symptom(2min post Definity®)

SECONDARY OUTCOMES:
Left Ventricular Opacification (LVO) | Day of Study
  The null hypothesis for efficacy (H0) will be: MVT-100 is not as effective as DEFINITY®. The alternative hypothesis (HA) for efficacy will be: MVT-100 is equivalently or more effective than DEFINITY®. Specifically, the following hypotheses will be tested:
  HA: LVO(MVT-100) ≥ LVO(Definity®) HA: SegmentVisualization(MVT-100) ≥ SegmentVisualization(Definity®)
Cardiac Segment Visualization | Day of Study
  The null hypothesis for efficacy (H0) will be: MVT-100 is not as effective as DEFINITY®. The alternative hypothesis (HA) for efficacy will be: MVT-100 is equivalently or more effective than DEFINITY®. Specifically, the following hypotheses will be tested:
  HA: LVO(MVT-100) ≥ LVO(Definity®) HA: SegmentVisualization(MVT-100) ≥ SegmentVisualization(Definity®)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith-Bindman R, Miglioretti DL, Johnson E, Lee C, Feigelson HS, Flynn M, Greenlee RT, Kruger RL, Hornbrook MC, Roblin D, Solberg LI, Vanneman N, Weinmann S, Williams AE. Use of diagnostic imaging studies and associated radiation exposure for patients enrolled in large integrated health care systems, 1996-2010. JAMA. 2012 Jun 13;307(22):2400-9. doi: 10.1001/jama.2012.5960. PMID 22692172
- [Background] Platts DG, Luis SA, Roper D, Burstow D, Call T, Forshaw A, Pascoe R. The safety profile of perflutren microsphere contrast echocardiography during rest and stress imaging: results from an Australian multicentre cohort. Heart Lung Circ. 2013 Dec;22(12):996-1002. doi: 10.1016/j.hlc.2013.05.637. Epub 2013 Jun 10. PMID 23764145
- [Background] Weissman, Neil J., Warren J. Manning, and Brian C. Downey. Contrast echocardiography: clinical applications. Waltham, MA : UpToDate, 2013.
- [Background] Lantheus Medical Imaging. Definity Package Insert. Definity Imaging. [Online] http://www.definityimaging.com/pdf/DEFINITY_US_PI_515987-0117.pdf.
- [Background] Pellikka PA, Nagueh SF, Elhendy AA, Kuehl CA, Sawada SG; American Society of Echocardiography. American Society of Echocardiography recommendations for performance, interpretation, and application of stress echocardiography. J Am Soc Echocardiogr. 2007 Sep;20(9):1021-41. doi: 10.1016/j.echo.2007.07.003. No abstract available. PMID 17765820
- [Background] Porter TR, Abdelmoneim S, Belcik JT, McCulloch ML, Mulvagh SL, Olson JJ, Porcelli C, Tsutsui JM, Wei K. Guidelines for the cardiac sonographer in the performance of contrast echocardiography: a focused update from the American Society of Echocardiography. J Am Soc Echocardiogr. 2014 Aug;27(8):797-810. doi: 10.1016/j.echo.2014.05.011. No abstract available. PMID 25085408